CLINICAL TRIAL: NCT01075035
Title: Evidence Based Multimodal Neurodiagnostic Imaging of Traumatic Brain Injury and Post-Traumatic Stress Disorder at the Saint Louis University Advanced Neurosurgical Innovation Center (SANIC)
Brief Title: Multimodal Neurodiagnostic Imaging of Traumatic Brain Injury and Post-Traumatic Stress Disorder
Acronym: SANIC
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: PT075832-R01; A-15194 (Other Grant/Funding Number: Department of Defense Study Number); IRB # 15919 (Other: SLU IRB #)
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2014-04

CONDITIONS: Traumatic Brain Injury; Post-Traumatic Stress Disorder
Keywords: Traumatic Brain Injury; TBI; Military; Imaging; MEG; PET/CT; MRI; fMRI; DTI; SANIC; veteran
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Normal Healthy Controls: Individuals with no history of Traumatic Brain Injury.
- Civilian TBI: Civilians who have had a Traumatic Brain Injury
- Military TBI: Combat military veterans who have had a Traumatic Brain Injury

SUMMARY:
The purpose of this study is to determine whether the brains of persons with and without traumatic brain injury differ in a meaningful way when advanced technology images of the brain are taken using three newer technologies that visualize the brain using a combination of external/internal magnetic fields and radioactive tracers (molecules that emit detectable particles). The hope is that the results of this study will validate tools (help prove that diagnostic tools actually detect disease) for the diagnosis and treatment of traumatic brain injuries (TBI).

DETAILED DESCRIPTION:
'Normal' appearing brain is often not normal when imaged with advanced neuroimaging techniques. It has been advocated that a battery of neurological assessments (including MEG) be developed to assess mild traumatic brain injury (TBI) and studies have shown that somatosensory evoked fields in severe TBI can serve as a measure of cortical function in comatosed TBI patients. Functional neuroimaging techniques such as PET and fMRI may reveal abnormalities in areas considered 'normal' on traditional MRI. Most significantly, advanced functional neuroimaging may enable customized neurorehabilitation planning with more efficient use of resources.

The study aim is to compare healthy brains, civilian TBI brains, and combat-related TBI to identify correlations between abnormal imaging parameters with neurorehabilitation potential utilizing advanced neurological imaging.

The study hypothesis states Severity of Traumatic Brain Injury (TBI) and Post-traumatic Stress Disorders (PTSD) can be detected and quantified using a multimodal battery of neurodiagnostic imaging techniques (MEG, PET/CT, 3 Tesla-MRI w/ DTI and fMRI) and rehabilitation potential can be predicted in the post acute phase.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age and non-active duty
2. Either:

   1. Normal (no history of head injury) -OR-
   2. TBI (injury since Jan. 1, 2002)

Exclusion Criteria:

1. Incapable of informed consent or absence of legally authorized representative.
2. Incarcerated (or subject to court supervision).
3. Known allergy to protocol contrast/imaging agent (or pregnant and unable to receive agent)
4. MRI incompatible (i.e. implant, metal, > 300 lbs, severe claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50-60 Normal Healthy Controls 50-60 Civilian TBI 50-60 Military TBI
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2008-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Neurocognitive Testing (PET/CT, MEG, fMRI w/ DTI)results | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bucholz, M.D., Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

REFERENCES:
- See also: St. Louis University Home Page for the Traumatic Brain Injury Study — https://sites.google.com/a/slu.edu/traumatic-brain-injury-study/